CLINICAL TRIAL: NCT07180706
Title: To Evaluate the Safety and Efficacy of Histotripsy for the Symptom Relief of Inoperable Abdominal Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202504142DIPC
Record Dates: First submitted 2025-07-31; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Tumors
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- treatment inoperable abdominal tumors (Experimental)
  Interventions: Device: Histotripsy

INTERVENTIONS:
Device: Histotripsy — Histotripsy is a tumor ablation technique developed in recent years that allows for non-invasive treatment of solid tumors using High-Intensity Focused Ultrasound (HIFU). This method works by physically focusing ultrasound energy at a single point within biological tissue, creating a focal zone of high-power, low-frequency ultrasound that induces mechanical fragmentation (histotripsy) and cavitation effects, dissolving the tissue into fragments and destroying tumor cells. Under real-time ultrasound imaging guidance, various scanning treatment protocols are used to move the focal point throughout the treatment zone, effectively ablating the tumor tissue. The destroyed tumor tissue is gradually absorbed by the body. Since this technique does not require needle puncture, electrode insertion, radiation, or thermal effects, it is minimally invasive and holds the potential to overcome the limitations of existing ablation technologies.

SUMMARY:
When solid tumors cause pain or other symptoms due to compression or mass effect, and surgical resection is not feasible, the primary clinical recommendation for malignant tumors is chemotherapy or local radiotherapy to delay tumor progression, improve quality of life, and prolong survival. For benign tumors, however, there are no other effective treatment options.

For unresectable tumors, local ablation techniques such as Radiofrequency Ablation (RFA) are considered as potentially curative alternatives. However, the main drawback of RFA is its invasive nature, which may sometimes cause bleeding or tumor seeding along the needle tract. Moreover, when tumors are adjacent to blood vessels, the efficacy of ablation is often compromised. Therefore, its application is currently limited mainly to small liver cancers.

Histotripsy is an emerging tumor ablation technology that utilizes High-Intensity Focused Ultrasound (HIFU) for non-invasive treatment of solid tumors. The mechanism involves physically focusing ultrasound energy to a precise location within biological tissue, where high-power and low-frequency ultrasound creates mechanical disruption (histotripsy) and cavitation effects to fragment the tissue and destroy tumor cells. Under real-time ultrasound imaging guidance and using multiple appropriate scanning strategies, the focal point moves within the treatment area to ablate tumor tissue. The destroyed tumor tissue is gradually absorbed by the body. Since this method does not require needle insertion or electrode placement and does not involve radiation or thermal injury, it is considered non-invasive and holds the potential to overcome current limitations of ablation techniques.

This clinical trial utilizes the Edison System developed by HistoSonics Inc., USA. The technology underwent its first multicenter Phase I human trial in 2018, treating 11 patients with advanced, multifocal liver tumors who were ineligible for surgical resection. All targeted liver tumors were successfully ablated with no device-related adverse events. Based on these results, a global multicenter, single-arm, non-randomized prospective trial (HOP4LIVER trial) was initiated in 2021 to assess the efficacy and safety of this system in treating primary and metastatic liver tumors. Imaging was conducted within 36 hours post-treatment to confirm technical success, and patients were monitored for 30 days, during which only three treatment-related adverse events occurred. A six-month post-operative evaluation showed a success rate of 95.5%. Consequently, the system received FDA De Novo approval in October 2023.

According to the HOPE4LIVER clinical trial, this treatment has demonstrated significant efficacy across various cancer types, including colorectal cancer with intrahepatic metastases (38%), pancreatic cancer (19%), and breast cancer (15%). Other cases included melanoma, neuroendocrine tumors, lung cancer, hemangiopericytoma, ovarian cancer, and bronchial cancer, indicating the potential applicability of this technique for other tumor types.

As the system has not yet been registered or approved by the Taiwan Ministry of Health and Welfare, investigators propose a research project targeting patients with intra-abdominal benign or malignant tumors who are unsuitable for surgical resection and are experiencing tumor-related symptoms. investigators aim to apply HIFU histotripsy for tumor ablation, monitor for any post-operative complications and symptom relief, assess tumor response after one month, and follow up on survival rates to evaluate the clinical feasibility and safety of this system.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years and older
* Diagnosed with a malignant liver tumor at National Taiwan University Hospital. - participants with intra-abdominal tumors measuring between 3 to 10 cm in diameter, such as hepatobiliary or pancreatic cancer, benign or malignant retroperitoneal tumors, or malignant sarcomas, who are experiencing tumor-related symptoms and discomfort.
* unresectable areas due to the presence of distant metastases, invasion of blood vessels or vital organs, or the risk of organ dysfunction resulting from tumor resection.
* participants with good physical condition, having an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1, and an American Society of Anesthesiologists (ASA) score of less than 3.
* No severe hepatic or renal dysfunction (Child-Pugh class A/B); total serum bilirubin ≤ 5 mg/dL; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within five times the upper limit of normal; serum creatinine within two times the upper limit of normal.
* Normal coagulation function, with a prothrombin time international normalized ratio (PT-INR) ≤ 2.0 and a platelet count above 100,000.
* Estimated life expectancy of more than three months.
* The maximum depth from the tumor to the skin surface is within 14 cm.

Exclusion Criteria:

* Tumors that cannot be clearly localized by ultrasound.
* Inability to find a safe internal path for ultrasound to reach the tumor during imaging evaluation, such as the presence of unsuitable media for ultrasound propagation like skin scars, intestinal gas, calcified tumors, and bones in the path.
* Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* Received treatment with an investigational agent/ procedure within 30 days prior to Histotripsy treatment
* Have undergone radiation therapy in the focused ultrasound treatment area within 30 days before or after treatment.
* arterial calcification in the ultrasound treatment area.
* Investigator-assessed contraindications
* Inability to undergo CT/MRI imaging
* Known history of HIV infection
* Tumor not clearly visualized on ultrasound
* No safe ultrasound pathway due to scarring, bowel gas, calcified tumor, or bone interference
* Prior radiotherapy within 30 days before or after treatment
* Arterial calcification in the treatment area
* arterial calcification in the ultrasound treatment area.
* Severe anesthesia intolerance
* Tumor invasion of major vessels, gastrointestinal tract, or respiratory tract
* within systemic infections; tissue ablation is not suitable until the infection is controlled.
* Other contraindications related to the medical device in this trial:

  1. Poor tolerance to anesthetics.
  2. The target tumor is less than 1 cm from the skin.
  3. within severe organ dysfunction, such as heart, liver, kidney, brain, or lung.
  4. within severe cachexia, extreme fatigue, or severe ascites.
  5. within severe diabetes.
  6. The treatment target involves important blood vessels or portal vein thrombosis, or the tumor has invaded the vessel wall or significantly compressed blood vessels.
  7. The tumor has invaded the digestive tract or respiratory tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
SF-36 with preoperative baseline within six months | six months
  The main goals are to confirm if the quality of life of subjects improves after treatment with a focused ultrasound system and to assess the safety of the treatment. SF-36 score range from 0 to 100, with higher scores indicating better health and
VAS with preoperative baseline within six months | six months
  The main goals are to confirm if the quality of life of subjects improves after treatment with a focused ultrasound system and to assess the safety of the treatment. VAS score measures pain intensity using a 10-cm line with "no pain" at 0 point and "worst possible pain" at 10 points.

SECONDARY OUTCOMES:
Comparison of Tumor Volume Before and After Treatment | seven months
  Comparison of tumor volume changes before and after treatment with the focused ultrasound system using CT/MRI imaging, based on RECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan